CLINICAL TRIAL: NCT01285765
Title: Randomized Phase III Study Evaluating the Non-inferiority of a Treatment Adapted to the Early Response Evaluated With 18F-FDG PET Compared to a Standard Treatment, for Patients Aged From 18 to 80 Years With Low Risk (aa IPI = 0) Diffuse Large B-cells Non Hodgkin's Lymphoma CD 20+
Brief Title: Evaluate a Treatment Adapted to the PET Response Compared to a Standard Treatment, for Low Risk DLBCL CD 20+ Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNH 2009-1B
Record Dates: First submitted 2011-01-14; First posted 2011-01-28 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: DLBCL

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-PET-result-adapted treatment (Experimental): 4 to 6 RCHOP21
  Interventions: Drug: RCHOP21
- standard treatment (Active Comparator): 6 RCHOP21
  Interventions: Drug: RCHOP21

INTERVENTIONS:
Drug: RCHOP21 — Prednisone-60 mg/m2: D1 D2 D3 D4 D5;Rituximab-375 mg/m2 : D1; Doxorubicin-50 mg/m2 D1;Cyclophosphamide-750 mg/m2:D1 Vincristine-1.4 mg/m2 :D1; G-CSF SC -5 microg/kg/day: D6 to D13
  Other Names: Rituximab-CHOP21

SUMMARY:
In this study, the investigators purpose is to evaluate the adaptation of treatment with early response based on PET scan results after 2 cycles of chemotherapy, for patient aged from 18 to 80 years, with low IPI DLBCL.

This is an open randomized study.

The primary endpoint is to evaluate the 3 years PFS with the aim to demonstrate the non inferiority of the experimental arm in comparison to standard arm:

In standard arm, the patients will receive 6 cycles of R-CHOP 21 without taking into account of PET scan results after 2 cycles.

In experimental arm, early good responder patients (defined as having a negative PET scan after 2 cycles, confirmed after 4 cycles) will receive only 4 cycles of R-CHOP 21.

In both arms, if the PET scan remains positive after 4 cycles of chemotherapy, a biopsy exam is needed to confirm the failure and an intensive chemotherapy is then recommended.

All of the patients, in both arms, will have an early evaluation with PET scan. All PET scan will be reviewed by a group of expert according to Deauville criteria defined by Meignan et al to adapt the decision after the 2nd cycle in experimental arm and after the 4th cycle for all patients. The final evaluation of response will be made according to 2007 Cheson's criteria.

DETAILED DESCRIPTION:
Localized stages DLBCL with low IPI (aaIPI = 0) have a very good prognostic after a standard immuno-chemotherapy with 6 cycles of R-CHOP 21. Five years PFS is estimated over 75%, whatever the age of the patient.

PET scan is actually considered as "the gold standard" for the initial staging and the evaluation of response after treatment. With this new technique, the response criteria have been redefined by Cheson and al. in 2007. Moreover, several recent studies showed that early evaluation of response with PET scan after only 2 cycles of chemotherapy was accurate to define two groups of patients:

"Early-good-responders", when PET scan is negative "Early-poor-responders", when PET scan remains positive Prognostic for the first group is very good, and for the second poorer. At the present time, the interest of the modification and/or the intensification of the treatment for the early-poor-responder patients is not demonstrated by any publication. New studies are ongoing for patients with advanced stages of DLBC NHL (GELA trial LNH 07-3B) or Hodgkin's lymphoma (GELA and EORTC trial H10); the aim is to evaluate a new strategy of treatment adapted to early response criteria.

No trial has already been made for low IPI DLBCL. In this study, the investigators purpose is to evaluate the adaptation of treatment with early response based on PET scan results after 2 cycles of chemotherapy, for patient aged from 18 to 80 years, with low IPI DLBCL.

This is an open randomized study.

The primary endpoint is to evaluate the 3 years PFS with the aim to demonstrate the non inferiority of the experimental arm in comparison to standard arm:

In standard arm, the patients will receive 6 cycles of R-CHOP 21 without taking into account of PET scan results after 2 cycles.

In experimental arm, early good responder patients (defined as having a negative PET scan after 2 cycles, confirmed after 4 cycles) will receive only 4 cycles of R-CHOP 21.

In both arms, if the PET scan remains positive after 4 cycles of chemotherapy, a biopsy exam is needed to confirm the failure and an intensive chemotherapy is then recommended.

All of the patients, in both arms, will have an early evaluation with PET scan. All PET scan will be reviewed by a group of expert according to Deauville criteria defined by Meignan et al to adapt the decision after the 2nd cycle in experimental arm and after the 4th cycle for all patients. The final evaluation of response will be made according to 2007 Cheson's criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven CD20+ diffuse large B-cell lymphoma (DLBCL) (WHO classification 2008) including clinical subtypes (primitive mediastinal, intravascular, etc.). Patients with De Novo Transformed DLBCL from low grade lymphoma (Follicular, other...) may also be included; or CD20+ B-cell lymphoma with intermediate features between DLBCL and Burkitt; or with intermediate features between DLBCL and classical Hodgkin lymphoma; or CD20+ Follicular lymphoma grade 3B; or CD20+ Aggressive B-cell lymphoma unclassifiable.
* Age from18 to 80 years.
* Patient not previously treated.
* Ann Arbor Stage : I or II.
* Normal level of LDH.
* ECOG performance status (PS) < 2.
* Age-adjusted international prognostic index (aaIPI) = 0.
* Baseline PET (PET0) performed before any treatment, even in absence of known lesion (for stage I for which the lesion has been removed for diagnostic reason).
* Having previously signed a written informed consent.
* The subject must be covered by a social security system (in France).

Exclusion Criteria:

* Any other histological type of lymphoma, Burkitt included.
* Any history of treated or non-treated small B-cell lymphoma.
* Central nervous system or meningeal involvement by lymphoma.
* Contra-indication to any drug contained in the chemotherapy regimens.
* Poor renal function (creatinin level >150 mmol/L), poor hepatic function (total bilirubin level >30 mmol/L, transaminases >2.5 ULN) unless these abnormalities are related to the lymphoma.
* Poor bone marrow reserve as defined by Absolute Neutrophils Count (ANC) <1.5 G/L or platelets <100 G/L, unless related to bone marrow infiltration.
* Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Any serious active disease (according to the investigator's decision).
* Positive HIV, HBV and HCV serologies before inclusion (except after hepatitis B vaccination or for patients who are HBs Ag negative, anti-HBs positive and/or anti-HBc positive but viral DNA negative).
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy.
* Pregnant or lactating women or women of childbearing potential not currently practicing an adequate method of contraception.
* Adult patient under tutelage.
* Impossibility to perform a baseline PET scan (PET0) before randomization and treatment start.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2020-05-23 (Actual); Study Completion 2020-05-23 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 3 years
  Evaluate by PFS at 3 years the non-inferiority of a chemotherapy treatment with 4 or 6 cycles of R-CHOP 21, determined according to early response assessed by PET at the end of 2 cycles versus standard chemotherapy of 6 cycles of R-CHOP 21 in patients with DLBCL lymphoma CD20+ with no factors of the IPI age adjusted.

SECONDARY OUTCOMES:
DELTA SUV | 3 weeks post C4 last patient
  Determine the decrease of SUV max between PET at baseline, PET after cycle 2 and PET after cycle 4 and evaluate the changes predictive interest.
Overall Survival, EFS, response duration, DFS | 3 years
  Assess the overall survival, the EFS (Event Free Survival - events defined as death from any cause, relapse for complete responders and undocumented complete responders, progression during or after treatment, initiation of a new anti-lymphoma therapy), the response duration, and the DFS for complete responders (disease free survival).
prognostic impact of the existence of a high tumor burden at diagnosis (> 10 cm) on PFS | 3 years
  Evaluate the prognostic impact of the existence of a high tumor burden at diagnosis (> 10 cm).
biological factors | 3 weeks post last cycle and 3years survival
  Identify the biological factors on blood samples and on tumor biopsy influencing the patient treatment response and prognosis.
Overall Response Rate | 3 weeks post last cycle last patient
  Evaluate the overall response rate according to IWC (International Harmonization Project - Cheson 2007) (CR, PR) after 4 or 6 cycles of R-CHOP21 according to the treatment arm.
Rate of good responders according to results at PET after C2 | 3 weeks post C2 last patient
  Evaluate the rate of negative PET2

CONTACTS AND LOCATIONS:
Overall Officials: Serge Bologna, MD, Principal Investigator — Centre d'Oncologie de Gentilly - Nancy - France; Jean-Noël BASTIE, MD, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (83):
- Belgium (14):
  - ZNA Stuivenberg, Antwerp
  - A. Z. Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - Université Catholique de Louvain Saint Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - UZ Gent, Ghent
  - Hôpital Jolimont, Haine-Saint-Paul
  - CHU de Liège, Liège
  - Clinique Saint Joseph, Mons
  - Clinique Saint Pierre, Ottignies
  - Centre Hospitalier de Wallonie Picarde - CHwapi, Tournai
  - CH de la Tourelle-Peltzer, Verviers
  - UCL Mont Godinne, Yvoir
- France (69):
  - CHU Angers, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - CH d'ARRAS, Arras
  - CH d'Avignon, Avignon
  - CH de la Côte Basque, Bayonne
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié - Bordeaux, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH du Dr Duchenne, Boulogne-sur-Mer
  - CH de Bourg-en-Bresse, Bourg-en-Bresse
  - IHBN - CHU Côte de Nacre, Caen
  - CH de Cannes, Cannes
  - Médipôle de Savoie, Challes-les-Eaux
  - Hôpital de Chalon, Chalon-sur-Saône
  - CH de Chambéry, Chambéry
  - Hôpital d'Instruction des Armées Percy, Clamart
  - CHU Estaing - Clermont Ferrand, Clermont-Ferrand
  - Hôpital Pasteur, Colmar
  - CH de Compiègne, Compiègne
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - CH Sud Francilien, Corbeil-Essonnes
  - Hôpital Henri MONDOR, Créteil
  - Chu Dijon, Dijon
  - CH de Dunkerque, Dunkirk
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
  - CH Départemental Vendée, La Roche-sur-Yon
  - CH de Versailles, Le Chesnay
  - CHU Bicetre, Le Kremlin-Bicêtre
  - CH de Lens, Lens
  - Hôpital Saint Vincent, Lille
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - Clinique Mutualiste Eugène André, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital des Chanaux, Mâcon
  - CH de Meaux, Meaux
  - CH Marc Jacquet, Melun
  - Hôpital Notre Dame du Bon Secours, Metz
  - CH de Mulhouse, Mulhouse
  - Centre d'Oncologie de Gentilly, Nancy
  - Centre Antoine Lacassagne, Nice
  - CHU de Nice, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital Saint Antoine, Service d'hématologie du Pr Marie, Paris
  - Hôpital Saint Antoine, Paris
  - Institut Curie, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - Hôpital Necker, Paris
  - Hôpital LYON SUD, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CH Rene Dubos, Pontoise
  - CH de la Région d'Annecy, Pringy
  - CHU de Reims, Reims
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Centre Hospitalier de Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - CH de Saint-Brieuc - Hôpital Yves Le Foll, Saint-Brieuc
  - Hôpital René Huguenin, Saint-Cloud
  - Institut de cancérologie de la Loire, Saint-Priest-en-Jarez
  - CHU de Strasbourg, Strasbourg
  - Hôpitaux du Leman, Thonon-les-Bains
  - Hôpital Sainte Musse, Toulon
  - CHU de Tours - Hôpital Bretonneau, Tours
  - CH de Troyes, Troyes
  - CH de Valence, Valence
  - CHU Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michot JM, Bologna S, Bastie JN, Borght TV, Briere J, Ribrag V, Bommier C, Peyrade F, Lebras L, Damaj G, Coso D, Sibon D, Bonnet C, Morschhauser F, Ghesquieres H, Fruchart C, Soussain C, Becker S, Olivier P, Julian A, Molina T, Haioun C, Tilly H. Early Positron Emission Tomography Response-Adapted Treatment in Low-Risk Diffuse Large B-Cell lymphoma: an open label, multicenter, randomised, non-inferiority phase 3 trial. Ann Oncol. 2025 Nov 17:S0923-7534(25)06264-7. doi: 10.1016/j.annonc.2025.11.006. Online ahead of print. PMID 41260259